CLINICAL TRIAL: NCT01161368
Title: A Phase II Study Evaluating the Efficacy and Safety of Lapatinib + Vinorelbine in ErbB2 Positive Metastatic Breast Cancer Patients Pretreated With Chemotherapy or Hormonal Treatment in Combination With Lapatinib for Metastatic Disease
Brief Title: A Study Evaluating the Efficacy and Safety of Lapatinib + Vinorelbine in ErbB2 Positive Metastatic Breast Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/BC.1.2.001
Record Dates: First submitted 2010-05-27; First posted 2010-07-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2014-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lapatinib, vinorelbine (Experimental): Drug: Lapatinib, Vinorelbine Lapatinib 1250mg orally once daily continuously
  plus
  Vinorelbine 20 mg/m2 intravenously (IV) once weekly [Days 1 and 8] for 2 weeks, followed by a rest week in a 3-week cycle.
  Interventions: Drug: Lapatinib, Vinorelbine

INTERVENTIONS:
Drug: Lapatinib, Vinorelbine — Lapatinib 1250mg orally once daily continuously
  plus
  Vinorelbine 20 mg/m2 intravenously (IV) once weekly [Days 1 and 8] for 2 weeks, followed by a rest week in a 3-week cycle.

SUMMARY:
The objective of this phase II study is to gain first information on the efficacy (PFS, ORR and OS) and safety of lapatinib plus vinorelbine in patients with HER2 positive metastatic breast cancer pretreated with a combination therapy (chemotherapy and/or hormonal therapy) including lapatinib and presenting with tumor progression.

Primary objective is to assess the efficacy with respect to the percentage of patients surviving without disease progression as assessed by RECIST criteria.

Secondary objectives are to assess the efficacy of the study treatment with respect to the objective response rates as assessed by RECIST criteria version 1.1, the overall survival and to evaluate the safety profile of the combination by recording the adverse events and abnormal laboratory values associated with the study treatments.

The main efficacy endpoints will be investigated both for the intent-to-treat (ITT) population and the per-protocol (PP) population.

DETAILED DESCRIPTION:
The objective of this phase II study is to gain first information on the efficacy (PFS, ORR and OS) and safety of lapatinib plus vinorelbine in patients with HER2 positive breast cancer pretreated with a combination therapy (chemotherapy, hormonal therapy) including lapatinib for metastatic disease.

The sample size is not based on statistical consideration. Thirty 30 patients are considered appropriate for a phase II study to gain first information on the efficacy and safety of the study treatment in the study indication.

Only descriptive statistical methods will be used to summarize the study results. Kaplan-Meier estimates will be calculated for PFS and OS. Median PFS and OS time and corresponding two sided 95% confidence intervals will be provided.

Categorical endpoints will be summarized in frequency tables and 95% confidence intervals will be calculated for the objective response rate (ORR) using RECIST.

All safety variables will be summarized descriptively The incidence of adverse events will be summarized by MedDRA terms in a descriptive manner.

The progression free survival time (PFS) is the primary efficacy endpoint of the study. Secondary outcomes are overall survival (OS) and objective response rates (ORR) using RECIST.

Safety outcomes are adverse events, safety laboratory data, physical examinations, vital signs, LVEF, ECG data and ECOG performance status

Definitions:

The objective response rate is the rate of subjects with complete response (CR) or partial response (PR).

Progression-free survival:

The time to progression or death is defined as the time from study entry until the first observation of disease progression or death due to any cause (whichever occurred earlier). Only those death will be considered, which occurs within 84 days of the last tumor assessment or study entry (whichever is later).

If a patient has no progression before a clinical cut-off or the death date is beyond the above-mentioned time interval after last tumor assessment, time to progression/death is censored on the date of last tumor assessment or study entry (in case of no post-baseline tumor assessment).

Overall survival will be calculated from study entry until death. For patients lost to follow-up, data will be censored at the time the patient was last determined to be alive.

As efficacy data of vinorelbine plus lapatinib are not available so far and the current protocol is applied as 2nd or 3rd line therapy for metastatic disease an ORR from 30-40% and a median PFS from 4-6 months is expected.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-specific procedure.
* Females ≥18 years.
* Histologically or cytologically confirmed, HER2-positive (HER+++ or HER++ and FISH positive), adenocarcinoma of the breast with measurable locally recurrent or metastatic disease, who are candidates for chemotherapy. Locally recurrent disease must not be amenable to radiotherapy or resection with curative intent.
* Presence of at least one measurable lesion according to RECIST Criteria version 1.1. (target lesion(s) must not lie within an irradiated area)
* Able to comply with the protocol.
* Prior treatment with a combination therapy including lapatinib as first or second-line treatment for metastatic disease.
* ECOG performance status of 0-1.
* Life expectancy more than 12 weeks.
* Adequate left ventricular ejection function at baseline, defined as LVEF ≥ 50% by either echocardiogram or MUGA.
* Adequate hematological function
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Hemoglobin ≥ 9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function
* Total bilirubin ≤ 1.25 x upper normal limit (ULN)
* AST, ALT ≤ 3.0 x ULN
* Adequate renal function: Serum creatinine ≤ 1.25 x
* ULN or calculated creatinine clearance ≥ 50 mL/min

Exclusion Criteria:

* Concomitant hormonal therapy for locally recurrent or metastatic disease. Note: previous hormonal therapy is allowed for adjuvant, locally recurrent or metastatic breast cancer, but must have been discontinued at least 1 week prior to first study drug administration.
* Previous radiotherapy for the treatment of metastatic disease (unless given for the relief of metastatic bone pain and with the precautions mentioned below).Radiotherapy administered solely for the relief of metastatic bone pain is allowed prior to study entry, providing that
* not more than 30% of marrow-bearing bone was irradiated
* the last fraction of radiotherapy was administered ≥ 3 weeks prior to first dose of Lapatinib.
* Other primary tumors/hematologic malignancies within the last 5 years, except for adequately controlled limited basal cell carcinoma of the skin, or carcinoma in situ of the cervix.
* Pre-existing peripheral neuropathy NCI CTCAE grade > 2 at first study drug administration
* Evidence of spinal cord compression or current evidence of central nervous system (CNS) metastases. If suspected, the patient should be scanned by CT or magnetic resonance imaging (MRI) within 28 days prior to first study drug administration to rule out spinal / CNS metastases.
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* History or evidence upon physical/neurological examination of CNS disease unrelated to cancer, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).
* Active infection requiring i.v. antibiotics at first study drug administration.
* Pregnant or lactating females. Pregnancy test to be assessed within 7 days prior to study treatment start.
* Women of childbearing potential (< 2 years after the last menstruation) not using effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) during the study and for a period of 6 months following the last administration of study drug.
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry
* Current or recent (within 28 days of first study drug treatment) treatment with another investigational drug or participation in another investigational study
* Clinically significant malabsorption syndrome or inability to take oral medication.
* Psychiatric disability judged by the Investigator to be interfering with compliance for oral drug intake.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Progressive Free Survival | 4 years
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

SECONDARY OUTCOMES:
Objective Response Rate using RECIST (vers 1.1) | 4 years
  * assess the efficacy of the study treatment with respect to the objective response rates as assessed by RECIST criteria version 1.1 the overall survival
  * evaluate the safety profile of the combination by recording the adverse events and abnormal laboratory values associated with the study treatments.
Overall survival (OS) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Lang, MD, Principal Investigator — National Institute of Oncology Rath Gyorgy u. 7-9. 1122 Budapest
Locations (2):
- Dep. of Medicine I , Division of Oncology, Vienna, Austria
- National Institute of Oncology, Budapest, Hungary